CLINICAL TRIAL: NCT05128136
Title: A 3-month Pilot Crossover Study in 24 US Couples to Compare Adherence, Preference and Acceptability of 3 Non-medicated Silicone Intravaginal Rings (IVRs) of Different External Diameters, Each Used for 30 Days
Brief Title: A Crossover Study Evaluating 3 Non-medicated Silicone IVRs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Albert Einstein College of Medicine (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 957
Record Dates: First submitted 2021-10-20; First posted 2021-11-19 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hiv; Pregnancy Related
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Masking Description: We propose a randomized, open-label, parallel group, 3-way crossover study comparing adherence, preference and overall acceptability of 3 different-sized placebo IVRs (IVRs A, B and C) in 24 couples. At enrollment, each woman will be randomly assigned to 1 of 6 sequences of IVR use (A-B-C, A-C-B, etc.) and will use each of the 3 IVRs (A, B and C) for 30d per IVR (90d total).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silicone IVR 46mm external diameter (Experimental): Non-medicated 46 mm ring.
  Interventions: Device: Impact of ring size on adherence
- Silicone IVR 56mm external diameter (Experimental): Non-medicated 56mm ring.
  Interventions: Device: Impact of ring size on adherence
- Silicone IVR 66mm external diameter (Experimental): Non-medicated 66mm ring.
  Interventions: Device: Impact of ring size on adherence

INTERVENTIONS:
Device: Impact of ring size on adherence — The study design is a randomized, open-label, parallel group 3-way crossover study comparing adherence, preference and overall acceptability of 3 different-sized placebo IVRs (IVRs A, B and C) in 24 US couples. At enrollment, each couple will be randomly assigned to 1 of 6 sequences of IVR use: A-B-C, A-C-B, B-A-C, B-C-A, C-A-B or C-B-A. Each couple will use each of the 3 IVRs (IVRs A, B and C) for 30 days per IVR, 90 days total.

SUMMARY:
The overall aim of this study is to assess different external diameters of intravaginal rings (IVRs) for adherence, preference, and acceptability. To assess these domains, women in male-partnered relationships will use three different size IVRs.

DETAILED DESCRIPTION:
The study design is a randomized, open-label, parallel group 3-way crossover study comparing adherence, preference and overall acceptability of 3 different-sized placebo IVRs (IVRs A, B and C) in 24 US couples. At enrollment, each couple will be randomly assigned to 1 of 6 sequences of IVR use: A-B-C, A-C-B, B-A-C, B-C-A, C-A-B or C-B-A. Each couple will use each of the 3 IVRs (IVRs A, B and C) for 30 days per IVR, 90 days total. Each couple will participate for approximately 4 months, including screening. After providing written informed consent at screening, females and their male partners will be evaluated against the inclusion and exclusion criteria by providing their medical, contraceptive, and sexual history as well as undergoing a clinical exam. The exam will include a visual inspection of the genitalia (men) and a speculum exam (women). Potential participants will be recruited by Emory University (Atlanta, GA) and Einstein College of Medicine (Bronx, NY) by contacting prior research participants who've consented to be contacted for new studies; advertising; and distribution of flyers in the study communities. All recruitment materials will be approved by the relevant IRBs prior to use. After screening, women will have an additional 4 visits and their male partners will have 1 additional in-person visit for enrollment and 3 remote visits. Before and after using each IVR, women will have a pelvic exam. If women report symptoms during interim visits, they will have a pelvic exam and will restart IVR use based on the clinical judgement of the site investigator. After enrollment, men who report symptoms possibly related to IVR use will be asked to attend the clinic for an examination. Follow-up visits (in-person for women and remote for men) will include counseling on protocol adherence, contraception, HIV risk reduction counseling. Women will be shown how to use the IVR at Visit 1/Enrollment and will be able to practice ring insertion and removal at that first visit. At monthly visits, women will be examined to check that the IVR is in place.

ADHERENCE: The primary adherence measure will be assessed via daily SMS text messages to women in which they will report if the IVR was out of the vagina in the previous 24h and if so, for how long. At monthly visits, women will respond to a computer assisted self-interview (CASI) questionnaire asking them to rate their adherence in terms of how well they feel they adhered to the IVR instructions for use. They will also be asked to report in more detail about expulsions and removals and the context in which those happen; feeling the ring during daily activities and during sex; and any symptoms experienced in the previous month.

PREFERENCE: We will ask women and their male partners to choose the IVR they think they will prefer at baseline -- before using any IVRs -- and then ask them to state their preference after using all 3 IVRs. Preferences at baseline and endline, and between males and females within each couple, will be compared.

ACCEPTABILITY: Acceptability will be assessed via the monthly CASI interviews according to an adapted version of the Merkatz et al IVR acceptability model.

SAFETY: Safety will be assessed by recording AEs.

ELIGIBILITY:
Inclusion Criteria:

Females:

* Aged 18-40 years old, inclusive, at Screening based on self-report
* Sexually active, defined as having had penile-vaginal sex with a male partner at least four times per month (e.g. once a week), on average, in the three months before Screening
* In a mutually monogamous relationship with the same male partner for at least 6 months prior to Screening, based on self-report
* Male partner is eligible and consents to participation
* Healthy based on medical history and physical exam at Screening
* Currently using effective non-vaginal contraception for at least 3 months prior to screening, including injectable, oral contraception, contraceptive patch or sterilization (male or female) based on self-report
* HIV-negative per test at Screening
* Not pregnant per urine pregnancy test at Screening and Enrollment
* Negative for chlamydia, gonorrhea, trichomoniasis or urinary tract infection (UTI) at screening
* Symptomatic vulvovaginal candidiasis or bacterial vaginosis (BV) at Screening. (Participants who test positive at initial screening may be treated and rescreened after completing treatment).
* Competent to provide written informed consent based on Investigator's assessment
* Owns or has access to Smart phone per self-report
* Agrees to not participate in any other clinical research for the duration of this trial

Males:

* Aged at least 18 years old at Screening based on self-report
* Sexually active, defined as having had penile-vaginal sex with a female partner at least four times per month (e.g. once a week), on average, in the three months before Screening
* In a mutually monogamous relationship with the same female partner for at least 6 months prior to Screening, based on self-report
* Female partner is eligible and consents to participation
* Healthy based on medical history and physical exam, including visual inspection of genitalia at Screening
* HIV-negative per test at Screening
* Negative for chlamydia, gonorrhea, trichomoniasis per tests at Screening (per local standard of care) at Screening
* Competent to provide written informed consent based on investigator's assessment
* Owns or has access to a Smart phone, per self-report
* Agrees to not participate in any other clinical research for the duration of this trial

Exclusion Criteria:

Females:

* Known or suspected allergy to silicone, as reported by participant
* Positive pregnancy test at Screening or Enrollment based on urine hCG test
* Positive for HIV per test at Screening
* Presence of any clinically significant genital epithelial findings (e.g. abrasions, ulcerations, lacerations, or vesicles) suspicious of STIs at Screening or Enrollment
* Positive chlamydia, gonorrhea, or trichomoniasis test at Screening (or Enrollment)
* Current urinary complaints or diagnosed UTI at Screening (or Enrollment)
* Presence of genital abnormalities via visual exam with speculum that would contraindicate IVR use at Screening or Enrollment
* Significant uterine or vaginal prolapse, or urethral obstruction
* Recurrent vaginitis (three or more episodes within the prior year)
* Unexplained vaginal bleeding per self-report within the 3 months before Screening
* Currently breastfeeding per self-report
* Partial or complete hysterectomy per self-report
* Gynecological surgery in the 6 months prior to Screening per self-report
* Within 6 weeks post abortion or 6 months postpartum, per Self-report.
* Using vaginal contraception (diaphragm, female condom, spermicide, IVR)
* Abnormal finding on examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data.
* Any other condition the clinician feels would jeopardize the health and wellbeing of the participant after assessing the participant's potential eligibility for the study
* Unable to comply with study requirements, including but not limited to, attending all study visits and using the IVRs as directed.
* Currently participating in any other clinical research trial involving investigational or marketed products

Males:

* Known or suspected allergy to silicone, as reported by
* Positive test for HIV at Screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence | Up to 90 days
  To determine which of 3 non-medicated IVRs each used continuously for 30 days yields the highest adherence as measured by the proportion of women who are adherent to instructions for IVR use for each for ~30 days continuously, based on daily text messages
Preference | Up to 90 days
  To assess which of 3 non-medicated IVRs each used continuously for 30 days is preferred by women and their male partners based on self reported preference by completing a questionnaire during and by the end of the study. Women and male partners will be asked to state their preference for one of the 3 IVRs at the end of the study.

SECONDARY OUTCOMES:
Acceptability | Up to 90 days
  Participants will be asked to respond to a questionnaire measuring domains of acceptability at the end of using each of the 3 IVRs. Acceptability will be measured by the IVR acceptability measurement tool (IAMT). We will also explore the association between demographics, previous contraceptive use, parity, sexual/vaginal practices, and menses on acceptability. We will compare preferences between women and their male partners and we will compare actual preference at the end of the study with assumed preferences at baseline.
Collection of Adverse Events | Up to 90 days
  To evaluate and compare the safety of 3 nonmedicated silicone IVRs each used and continuously for 30 days as measured by the number and percent of participants with AEs and serious AEs. AEs will be summarized overall by severity and by relation to product use. AEs that are potentially related could be abrasion or erythema due to the device.
Patterns of adherence | 90 days
  To explore patterns of adherence based on frequency of removals and expulsions per IVR and overall; duration of removals and expulsions per IVR and overall; reasons for removals for each IVR and overall; activities associated with expulsions per IVR and overall; and association between demographics and other background characteristics, sexual activity, and menstruation on adherence to each IVR and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Friedland, MPH, Study Director — Population Council
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Albert Einstein College of Medicine,, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gottert A, Friedland BA, Plagianos M, Zieman B, Sales JM, Atrio J, Shetty S, Sant'Anna Marinho C, Roselli N, Merkatz R, Bruce I, Haddad LB. Development and Validation of a Multidimensional Intravaginal Ring Acceptability Scale Among US Women and Their Male Partners. Perspect Sex Reprod Health. 2025 Jun;57(2):144-153. doi: 10.1111/psrh.70009. Epub 2025 Apr 11. PMID 40211751